CLINICAL TRIAL: NCT06840834
Title: Assessment of Ivonescimab as Salvage Treatment in Relapsing Pleural Mesothelioma Patients, Previously Treated by Immunotherapy and Standard Chemotherapy
Brief Title: Evaluating Ivonescimab as a Potential Treatment for Pleural Mesothelioma Patients Whose Cancer Has Returned After Previous Immunotherapy and Chemotherapy
Acronym: Bi-MAPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2403; 2024-519052-82-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-05; First posted 2025-02-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pleural Mesotheliomas
Keywords: pleural mesothelioma; ivonescimab; bispecific antibody; anti-VEGF; anti-PD-1
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab (Experimental): 20 mg/kg IV (a fixed dose of 3200 mg for ivonescimab should be used for patients with weight ≥160 kg), every 3 weeks.
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab is administered IV Q3W on Day 1 of each cycle. Ivonescimab is given at a dose of 20 mg/kg (a fixed dose of 3200 mg for ivonescimab should be used for patients ≥160 kg). The total duration of ivonescimab treatment is up to 24 months.
  Other Names: SMT112

SUMMARY:
Multicentre, open-label, single arm phase II study for patients with PM previously treated by immunotherapy and standard chemotherapy. 38 patients will be given second or third-line treatment with ivonescimab 20mg/kg every 3 weeks.

An estimated 38 patients will be enrolled in approximately 20 centres. Patients will be treated for a maximum of 2 years, until disease progression, unacceptable toxicity, withdrawal of consent or another discontinuation criterion is met.

The null hypothesis is disease control rate (DCR) at 12 weeks ≤ 30%. The alternative hypothesis is DCR ≥ 55% at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent. Subjects must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

   Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Histologically-proven Pleural Mesothelioma (no cytology allowed, biopsies by thoracoscopy recommended).

   Note: pathology certification by national expert network NETMESO/MESOPATH should be checked as already done in routine in France by NETMESO regional expert MTB for PM (or similar national certification if the patient had his/her PM diagnosis obtained outside France, e.g. Belgium).
3. Documented progression by CT with iodine injection according to modified RECIST 1.1 for mesothelioma (mRECIST 1.1; pleural thickness perpendicular to the chest wall or mediastinum of 7mm or more, on 2 positions, at 3 separate levels on transverse cuts of CT-scan, at least 1cm apart, the sum of 6 measurements defining a pleural unidimensional measure), or according to RECIST 1.1 for mediastinal nodes or metastatic lesion, after maximum 2 lines including immunotherapy by nivolumab ± ipilimumab, and standard P/P chemotherapy [with (maximum 40% total of patients) or without bevacizumab], sequentially (regardless of treatment order), or first-line combining standard chemotherapy + IO (pembrolizumab or other IO investigational drug but no anti-angiogenic drug).
4. Measurable disease according to mRECIST 1.1.
5. ECOG PS 0 or 1.
6. Weight loss <10% within 3 months of study entry.
7. Age ≥18 years.
8. Life expectancy >3 months.
9. Available pathological samples (at least 10 slides from the thoracoscopy biopsies) for centralized PD-L1, MTAP, immunohistochemistry, and NGS / transcriptome analyses, all slides being centrally reviewed by the French panel MESOPATH for mesothelioma histological certification. If archival tissue is either insufficient or unavailable, the patient may still be eligible upon discussion with IFCT.
10. Adequate biological functions:

    Creatinine Clearance ≥45 mL/min (Cockroft or MDRD or CKD-epi); neutrophils

    ≥1500/mm3; platelets ≥100 000/mm3; haemoglobin ≥9 g/dL; AST and ALT <3 x ULN, total bilirubin <2 x ULN (patients with hepatic metastases or Gilbert's syndrome must have AST and ALT ≤5 x ULN and a baseline total bilirubin ≤2 x ULN), urine protein <2+ or 24 hours urine protein quantification <1.0 g, prothrombin time (PT) or international normalized ratio (INR) ≤1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless abnormalities are unrelated to coagulopathy or are secondary to prophylactic coagulation).
11. Women of childbearing potential and sexually active should use a highly effective contraception method within the 28 days preceding the first dose and during the 6 months following the last dose of treatment. Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
12. For male subjects who are sexually active with women of childbearing potential, an efficacious contraception method should be used during the treatment and during the 6 months following the last dose.
13. Patient covered by a national health insurance.

Exclusion Criteria:

1. ECOG PS>1.
2. Previous treatment for PM by more than 2 lines of systemic treatment, or by bevacizumab (or another anti-angiogenic / anti-VEGF pathway drug) except if combined with P/P chemotherapy [scheme validated by ASCO, NCCN, and ESMO guidelines] in maximum 40% of the total of recruited patients (n=15).
3. Suspicion of hyperprogressive disease or rapid tumour progression when treated by previous IO (i.e. progressive disease within 9 weeks of treatment by previous nivolumab ± ipilimumab or alternative immunotherapy, starting from C1D1 or from randomization if previous experimental immunotherapy).
4. Pleural effusion as the only radiological abnormality without measurable pleural thickness or mediastinal node enlargement.
5. Peritoneal, pericardial or tunica vaginalis testis mesothelioma, without any pleural involvement at the time of diagnosis.
6. Previous diagnosis of adenocarcinoma from any anatomic site within the previous 3 years, with the exception of prostate adenocarcinoma history in case of localized prostate cancer with good prognostic factors according to d'Amico classification (<T2a, Gleason score ≤6 and PSA ≤10 ng/ml), provided they were treated in a curative modality (surgery or radiotherapy, without any chemotherapy).
7. Previous or active cancer within the previous 3 years (except for already treated in situ carcinoma of the cervix, or basal cell skin cancer, treated or not).
8. Uncontrolled pleural effusion despite previous (talc or other) pleurodesis, requiring thoracocentesis (by pleural aspiration) more often than every 21 days. However, patients with efficient indwelling pleural catheter (IPC) are eligible.
9. Symptomatic untreated brain metastasis (without previous whole brain radiotherapy or stereotactic ablative brain radiotherapy or without surgical resection). At least 2 weeks delay between the end of radiotherapy and the beginning of the treatment should be respected. Asymptomatic brain metastasis, not needing corticosteroids (>10 mg prednisone equivalent daily) or mannitol infusions, are allowed.
10. Radiotherapy needed at initiation of treatment, except bone palliative radiotherapy on a painful or compressive tumour site (in this case, target lesions should not be selected in the irradiated zone).
11. History of previous primary immunodeficiency, organ transplantation needing an immunosuppressive treatment, any immunosuppressive drug within 28 days before registration date, or history of severe toxicity (grade 3/4) by immune mechanism linked to another immunotherapy treatment for any kind of disease.
12. Systemic treatment with corticosteroids with a dose >10 mg prednisone equivalent daily, within 14 days before initiation of the treatment. Inhaled, nasal or topical corticosteroids are allowed.
13. History of active autoimmune disease, needing systemic immunosuppressive drug, including but not limited to rheumatoid polyarthritis, myasthenia, autoimmune hepatitis, systemic Lupus, Wegener's granulomatosis, vascular thrombosis associated with anti-phospholipid syndrome, Sjogren's syndrome with interstitial pulmonary disease, Guillain-Barré syndrome within previous 15 years, multiple sclerosis, vasculitis, or glomerulonephritis.

    Patients with type I diabetes, or hypothyroidism, or immune cutaneous disease (vitiligo, psoriasis, alopecia) or benign rheumatoid polyarthritis not needing any immunosuppressive systemic treatment or >10 mg daily oral steroids, or benign sicca syndrome (Sjogren) without interstitial lung disease (ILD), or history of past Guillain-Barre syndrome beyond 15 previous years, totally reversible with no sequelae, no systemic immunosuppressive treatment during the last 20 years, are allowed to be included. Patients with Grave's disease or psoriasis not requiring systemic therapy within the previous two years from are allowed to be included.
14. Active inflammatory intestinal disease (diverticulosis, Crohn's disease, haemorrhagic recto-colitis, coeliac disease) or any serious chronic intestinal disease with uncontrolled diarrhoea.
15. Pre-existing moderate or severe ILD as assessed by the diagnostic CT-scan and decrease of TLCO higher than 35% from theoretical normal values linked to such ILD.
16. Major surgical procedures or serious trauma within 4 weeks prior to inclusion or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to registration.
17. History of bleeding tendencies or coagulopathy, or clinically significant bleeding symptoms or risk within 4 weeks prior to inclusion, including but not limited to: gastrointestinal bleeding; haemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots), note: transient haemoptysis associated with diagnostic bronchoscopy is allowed; nasal bleeding / epistaxis (bloody nasal discharge is allowed); need for therapeutic anticoagulant therapy within 14 days prior to inclusion. Note: prophylactic anticoagulation for deep vein thrombosis / pulmonary embolism or to maintain venous patency is allowed.
18. Current hypertension with systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive therapy.
19. History of major diseases before registration, specifically:

    1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or vascular disease (e.g. aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to inclusion, or other cardiac impairment that may affect the safety evaluation of the study drug (e.g. poorly controlled arrhythmias, myocardial ischemia). Patients with a significant cardiac history, even if controlled, should have a LVEF >45%.
    2. History of oesophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses or acute gastrointestinal bleeding within 6 months before inclusion.
    3. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to inclusion.
    4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks prior to inclusion.
    5. History of perforation of the gastrointestinal tract or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to inclusion.
20. Imaging during the screening period shows that the patient has:

    1. Radiologically documented evidence of major lung blood vessel invasion or encasement by cancer.
    2. Radiographic evidence of lung intratumor cavitation.
21. Active uncontrolled infection including active tuberculosis, known acute viral hepatitis B and C according to serological tests. Patients with serological sequelae of cured viral hepatitis are allowed to be included. Past primary pulmonary tuberculosis in youth does not consist of a contra-indication. Past tuberculosis disease history does not represent a contraindication provided the patient was treated for at least 6 months by anti-tuberculosis antibiotic treatment.
22. Patients with a known history of a positive test for HIV or known AIDS who have not received effective antiretroviral therapy (ART) for the last 4 weeks and who have an HIV viral load >200 copies/mL, regardless of CD4+ T-cell count.
23. Living attenuated vaccine received within the 30 previous days; mRNA and adenovirus vector anti-SARS-CoV2 vaccine are allowed.
24. Inability to comply with study or follow-up procedures as estimated by the referent investigator.
25. Known allergy or hypersensitivity to study treatment or any excipient.
26. Concomitant treatment with another experimental treatment or participation in another clinical trial.
27. Patient who is subject to legal protection or who is unable to express his will.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the therapeutic value of the bispecific antibody anti-VEGF / anti-PD-1 ivonescimab as 2nd/3rd line treatment in relapsing PM patients | 12 weeks after start of treatment.
  The analysis of the primary efficacy endpoint will be conducted in all eligible patients, based on the disease control rate (DCR) at 12 weeks according to mRECIST 1.1 for mesothelioma, which was defined as the proportion of patients with compete response (CR), partial response (PR) or stable disease (SD) at 12 weeks as assessed by the independent review committtee.

SECONDARY OUTCOMES:
Tolerance, safety of treatment | From time of informed consent through treatment period and up to 90 days post last dose of study treatment (maximum of 2 years and 3 months).
  Incidence, nature and severity of AEs, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0).
Progression free survival (PFS) | At progression, up to 2 years after start of treatment.
  PFS is defined as the time from date of inclusion to the earliest date of disease progression, as determined by Investigator review and review of radiographic disease assessments by IRC as per mRECIST v1.1 for mesothelioma, or death due to any cause. If a patient has not had a PFS event at the time of the analysis cut-off or at the start of any new anticancer therapy, PFS is censored at the date of last adequate tumour assessment.
Overall survival | Around 45 months.
  Overall survival is defined as the time from date of inclusion to the date of death due to any cause. If a death has not been observed by the date of the analysis cut-off, OS will be censored at the date of last contact.
Best response rate | At progression, up to 2 years after start of treatment.
  Best response rate is defined as the percentage of patients who have achieved a best response of a complete response (CR) or partial response (PR) as determined by Investigator review and review of radiographic disease assessments by IRC as per mRECIST v1.1 for mesothelioma.
Duration of response | At progression, up to 2 years after start of treatment.
  DOR is defined as the time from the date of the first response (CR or PR) to the earliest date of disease progression, as determined by Investigator review and review of radiographic disease assessments by IRC as per mRECIST v1.1 for mesothelioma, or death due to any cause. If a patient with a CR or PR has neither progressed nor died at the time of the analysis cut-off or at the start of any new anticancer therapy, the patient will be censored at the date of last adequate tumour assessment. DOR will be calculated for patients who have achieved a confirmed overall response (i.e. CR or PR).

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Besançon - CHU, Besançon
  - Brest - CHU, Brest
  - Caen - CHU, Caen
  - Clermont-Ferrand - Centre Jean Perrin, Clermont-Ferrand
  - Créteil - CHI, Créteil
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Lille - CHU, Lille
  - Marseille - APHM, Marseille
  - Montpellier - CHU, Montpellier
  - Mulhouse - GHRMSA, Mulhouse
  - Nantes - Hôpital Laennec, Nantes
  - Paris - Bichat, Paris
  - Bordeaux - CHU, Pessac
  - Lyon - HCL, Pierre-Bénite
  - Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Toulon - CHI, Toulon
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Metz - Hôpital Robert Schuman, Vantoux

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ifct.fr